CLINICAL TRIAL: NCT00482625
Title: Phase IIA Trial Testing Erlotinib as an Intervention Against Intraductal Pancreatic Mucinous Neoplasms
Brief Title: Erlotinib Hydrochloride in Treating Patients With Pancreatic Cancer That Can Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The protocol has been completed prematurely (e.g., due to poor accrual, insufficient drug supply, IND closure).
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00898; UCI 06-30; N01CN35160 (NIH); CDR0000547235 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-03

CONDITIONS: Intraductal Papillary Mucinous Neoplasm of the Pancreas; Recurrent Pancreatic Cancer; Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms; Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Surgical Procedures, Operative; Congresses as Topic; Immunohistochemistry; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive erlotinib hydrochloride PO QD for 21-42 days. Patients then proceed to surgery.
  Interventions: Drug: erlotinib hydrochloride; Procedure: conventional surgery; Other: immunohistochemistry staining method; Genetic: protein expression analysis; Procedure: biopsy; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Procedure: conventional surgery — Undergo pancreatectomy
  Other Names: surgery, conventional
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: protein expression analysis — Correlative studies
Procedure: biopsy — Correlative studies
  Other Names: biopsies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving erlotinib hydrochloride before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. This phase II trial is studying how well erlotinib hydrochloride works in treating patients with pancreatic cancer that can be removed by surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that the activated epidermal growth factor receptor (EGFR) signal transduction biomarker Mucin 5AC (MUC5AC) protein expression within intraductal pancreatic mucinous neoplasm (IPMN) lesions will have greater than zero absolute mean decrease from baseline comparing pre and post 21-42 days of Erlotinib (erlotinib hydrochloride) administration at 100mg orally (PO) once daily (QD).

SECONDARY OBJECTIVES:

I. To test the hypothesis that other correlative IPMN EGF inducible biomarkers will have greater than zero absolute mean decrease from baseline pre and post Erlotinib 100mg PO QD therapy.

II. Safety of Erlotinib treatment. III. To determine Erlotinib pharmacokinetic concentration in plasma and pancreatic tissue at the 100mg/day dose up to 42 days of therapy.

OUTLINE:

Patients receive erlotinib hydrochloride PO QD for 21-42 days in the absence of disease progression or unacceptable toxicity. Patients then undergo to pancreatectomy.

After completion of study treatment, patients are followed up at 4-20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed IPMN histological diagnosis, endoscopic ultrasound fine needle aspiration (EUS-FNA) core biopsy tissue specimen with plan for pancreatic surgical resection; histological diagnosis should be within 6 months of entry into protocol
* Patients must have adequate bone marrow function at study entry
* White blood cell (WBC) > 3,000
* Platelets > 100,000/mm^3
* Hemoglobin > 10 g/dL
* Plasma creatinine of < 1.6 mg/dL
* Total bilirubin < 1.5
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5 x upper limit of normal
* Patients with evidence of obstructive lung disease (forced expiratory volume in one second [FEV1] < 80% predicted and FEV1/forced vital capacity [FVC] ratio < 90% of predicted value) as the etiology of a low diffusing capacity will still be eligible as long as the chest radiograph or computed tomography (CT) does not demonstrate interstitial changes
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Women of child-bearing potential and men taking study drug must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand, as well as sign the written informed consent document
* If a woman of child-bearing potential, must have a negative pregnancy test prior to study entry; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately

Exclusion Criteria:

* Intake of EGFR antagonist, Erbitux (cetuximab)
* Previous history of sensitivity to Tarceva (erlotinib hydrochloride), Iressa (gefitinib), or Erbitux, such as a rash that is uncontrollable by topical steroids and/or antibiotics
* Uncontrollable diarrhea of any cause
* Active keratoconjunctivitis, or corneal surgery in the past three weeks
* Participants taking a known cytochrome P450 3A4 (CYP 3A4) inducer (e.g., phenytoin, carbamazepine, St. John's wort, and rifampin) and medications known to be inhibitors or metabolized by CYP3A4; these inhibitors include erythromycin, clarithromycin and ketoconazole, and patients taking them will be excluded since these drugs may be expected to result in altered exposure of Erlotinib
* Hospitalization within the past 5 years for mania or for bipolar disease
* Participants may not be receiving any other investigational pharmaceutical agents
* Women who are breast-feeding should not receive Erlotinib
* Any medical or psychosocial condition that, in the opinion of the investigator, could jeopardize the subject's participation in and compliance to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-06; Primary Completion 2010-02 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Lipkin, MD,PhD, Principal Investigator — Weill Cornell College of Medicine
Locations (1):
- University of California Medical Center At Irvine-Orange Campus, Orange, California, United States

REFERENCES:
- [Result] Armstrong WB, Wan XS, Kennedy AR, Taylor TH, Meyskens FL Jr. Development of the Bowman-Birk inhibitor for oral cancer chemoprevention and analysis of Neu immunohistochemical staining intensity with Bowman-Birk inhibitor concentrate treatment. Laryngoscope. 2003 Oct;113(10):1687-702. doi: 10.1097/00005537-200310000-00007. PMID 14520092

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.17 (14.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Number of Positive IPMN Celss and Staining Intensity After Treatment
Description: Number of participants showed a reduction in number of positive IPMN cells and staining intensity after treatment
Time Frame: Pre-treatment and post-treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 3
participants | 2

2. Secondary Outcome: Plasma Calculated Concentration - OSI-774 (ng/mL)
Description: Plasma concentration levels of Erlotinib (OSI-774)
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 4
ng/mL | 428.5 (290.4)

3. Secondary Outcome: Pancreas Calculated Concentration - OSI-774 (ng/g)
Description: Pancreatic tissue concentration levels of Erlotinib (OSI-774)
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 4
ng/g | 188.7 (121.7)

4. Secondary Outcome: Plasma Calculated Concentration - OSI-420 (ng/mL)
Description: Plasma concentration levels of Erlotinib (OSI-420)
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 4
ng/mL | 27.6 (21.3)

5. Secondary Outcome: Pancreas Calculated Concentration - OSI-420 (ng/g)
Description: Pancreatic tissue concentration levels of Erlotinib (OSI-420)
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 4
ng/g | 17.3 (7.2)

6. Secondary Outcome: Number of Participants Reported at Least 1 Adverse Event With a Grade of 3 and Above
Description: The worst grade of pre-listed toxicity will be summarized by participant and by visit for each treatment group. Descriptive statistics (frequencies and percents) will be used to summarize data and hypotheses about group differences will be tested where appropriate.
Time Frame: Up to 20 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 6
participants | 0

ADVERSE EVENTS:
Time Frame: All adverse events are reported and docuemted during the study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=6)
DIARRHEA (Gastrointestinal disorders) | 3 (3)
DIFFICULTY DIGESTING FOOD-UPPER GI (Gastrointestinal disorders) | 1 (1)
DRY EYES (Eye disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
DRY SKIN ON BODY (Skin and subcutaneous tissue disorders) | 1 (1)
DRY SKIN ON CHEEK AND CORNERS OF MOUTH (Skin and subcutaneous tissue disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
LEG, FOOT, ANKLE CRAMPS (Musculoskeletal and connective tissue disorders) | 1 (1)
LOSS OF APPETITE (Gastrointestinal disorders) | 1 (1)
OUT OF RANGE LYMPHOCYTE VALUE-CLINICALLY SIGNIFICANT (Investigations) | 1 (1)
OUT OF RANGE NEUTROPHIL VALUE-CLINICALLY SIGNIFICANT (Investigations) | 1 (1)
OUT OF RANGE WBC VALUE-CLINICALLY SIGNIFICANT (Investigations) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less